CLINICAL TRIAL: NCT00333398
Title: A Phase III, Randomized, Double-Blinded, Placebo-Controlled, Multi-Center Study to Evaluate the Immunogenicity, Safety and Tolerability of CSL Limited Inactivated Influenza Vaccine in Adults Greater Than or Equal to 18 to Less Than 65 Years of Age
Brief Title: Immunogenicity, Safety and Tolerability of CSL Limited Inactivated Influenza Vaccine in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 06-0016; CSL-CT-FLU-05-09
Record Dates: First submitted 2006-06-01; First posted 2006-06-05 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2008-06

CONDITIONS: Influenza
Keywords: CSL Influenza Vaccine, influenza, vaccine, immunogenicity
MeSH Terms: conditions — Influenza, Human | interventions — Thimerosal

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Experimental): 250 subjects-Lot #1 multiple-dose vial (thimerosal-containing).
  Interventions: Biological: CSL Trivalent Inactivated Influenza Vaccine with Thimerosal
- 2 (Experimental): 250 subjects-Lot #2 multiple-dose vial (thimerosal-containing).
  Interventions: Biological: CSL Trivalent Inactivated Influenza Vaccine with Thimerosal
- 3 (Experimental): 250 subjects-Lot #3 multiple-dose vial (thimerosal-containing).
  Interventions: Biological: CSL Trivalent Inactivated Influenza Vaccine with Thimerosal
- 4 (Placebo Comparator): 250 subjects-multiple-dose vial placebo (thimerosal-containing).
  Interventions: Biological: Placebo with Thimerosal
- 5 (Experimental): 250 subjects-Prefilled Lot #1, #2, or #3 (TBD) (thimerosal-free).
  Interventions: Biological: CSL Trivalent Inactivated Influenza Vaccine - Thimerosal-free

INTERVENTIONS:
Biological: CSL Trivalent Inactivated Influenza Vaccine - Thimerosal-free — CSL influenza vaccine-prefilled syringe presentation (thimerosal-free) 15 mcg per dose of each of the hemagglutinins of H1N1, H3N2, and B strains (total of 45 mcg of hemagglutinins). Single dose of 0.5 mL administered on study day 0.
  Arms: 5
Biological: CSL Trivalent Inactivated Influenza Vaccine with Thimerosal — CSL influenza vaccine-multiple dose vial presentation (thimerosal-containing) containing 15 mcg per dose of each of the hemagglutinins of H1N1, H3N2, and B strains (total of 45 mcg of hemagglutinins). Single dose of 0.5 mL administered on study day 0.
  Arms: 1; 2; 3
Biological: Placebo with Thimerosal — Phosphate buffered isotonic saline solution containing thimerosal. Single dose of 0.5 mL administered on study day 0.
  Arms: 4

SUMMARY:
The purpose of this study is to investigate the effectiveness, safety, and tolerability of an influenza vaccine. Influenza is a highly infectious disease that occurs throughout the world in the winter months. Infection with an influenza virus is a major public health threat as it has the ability to spread rapidly and affect large numbers of people. Up to 1359 healthy adults ages 18 to less than 65 years old will participate in this study for up to 24 days. Volunteers will receive an injection of either influenza vaccine with thimerosal, vaccine without thimerosal, or placebo with thimerosal. Volunteers will be asked to document information about any health changes for 21 days following vaccination. Volunteers will return to the clinic on days 5 and 21 after vaccination to share this information with study staff. On day 21, volunteers will have a physical examination. Blood samples will be taken prior to vaccination and at Day 21 post-vaccination.

DETAILED DESCRIPTION:
The purpose of this Phase III, randomized, double-blinded, placebo-controlled, multi-center study is to evaluate the immunogenicity, safety, and tolerability of CSL Limited Inactivated Influenza Vaccine in adults ages 18 to less than 65. The primary objective of this study is to demonstrate that vaccination with CSL Limited Inactivated Influenza Vaccine produces an immune response sufficient to meet the Committee for Medicinal Products for Human Use (CHMP) criteria for young adults of 40% serorconversion and 70% seroprotection. Secondary objectives are to: demonstrate clinical consistency between 3 lots (batches) of CSL Limited Inactivated Influenza Vaccine multi-dose vial presentation (Thimerosal containing); to demonstrate clinical consistency between CSL Limited Inactivated Influenza Vaccine multi-dose vial presentation (Thimerosal containing) and CSL Limited Inactivated Influenza Vaccine pre-filled syringe presentation (Thimerosal-free); and to demonstrate acceptable safety and tolerability of CSL Limited Inactivated Influenza Vaccine multi-dose vial presentation (Thimerosal containing) and pre-filled syringe presentation (Thimerosal-free). Primary endpoints are seroprotection rate and seroconversion rate. Seroprotection is defined as a minimum post-vaccination humagglutination inhibition (HI) titer of 1:40, and seroconversion is defined as an increase in HI antibody titer of at least 4-fold, with a minimum post-vaccination HI titer of 1:40. Secondary endpoints are: comparison of the Geometric Mean Titers to influenza hemagglutinin antigens post vaccination of the active treatment arms; and the number and rate of the type, frequency and intensity of adverse events (AE) in the active treatment arms. Approximately 1250 (and up to 1359) healthy adults, ages 18 to less than 65 years old, will be enrolled into this clinical trial. Subjects who meet the inclusion criteria for the study will be randomized in a 1:1:1:1:1 ratio to receive 1 of 3 lots of vaccine in multidose vials, a single lot of vaccine in pre-filled syringes or placebo in multi-dose vials (250 subjects per group). Vaccine will be prepared and administered by an unblinded vaccine administrator, who will not be involved in subsequent assessments. Subjects will be observed in the clinic for at least 30 minutes after vaccination, and subjects will maintain a 5-day, post-vaccination solicited AE and local reaction memory aid and a 21-day unsolicited AE memory aid. Subjects will return to the clinic at day 5 to review their reactogenicity memory aid. Subjects will also return to clinic on Day-21 post-vaccination for AE and concomitant medication assessment, a targeted physical examination (if indicated), and a review of the memory aid. Serum for antibody titers will be drawn prior to vaccination and on Day-21 post-vaccination. Subjects will participate for up to 24 days.

ELIGIBILITY:
Inclusion Criteria:

* Is a healthy male or nonpregnant female (as indicated by a negative urine or serum pregnancy test immediately prior to vaccine administration) aged greater than or equal to 18 years to less than 65 years at the time of informed consent.
* Provides written informed consent to participate in the study and adherence to all protocol requirements.
* Is in good health, as determined by vital signs (heart rate, blood pressure, oral temperature), medical history, and a targeted physical examination based on medical history.
* Is able to understand and comply with planned study procedures.
* Is female of nonchildbearing potential, ie, either surgically sterilized or 1 year postmenopausal. If female is of child bearing potential, she must be abstinent or using adequate contraceptive precautions, eg, intrauterine device, oral contraceptive, or equivalent hormonal contraception (eg, progestogen-only implant, cutaneous hormonal patch, injectable contraceptives, or diaphragm) and agree to continue such precautions for 2 months after vaccination.

Exclusion Criteria:

* Known hypersensitivity to a previous dose of influenza vaccine or allergy to eggs, chicken feathers, neomycin, polymyxin, thimerosal, or any components of the study vaccines.
* Has been vaccinated against influenza in the previous 6 months.
* Has underlying medical condition for which influenza vaccination is recommended; chronic heart or lung condition including asthma; metabolic disease; kidney disease; blood disorder (such as sickle cell anemia); or weakened immune system including HIV/AIDS.
* Has acute clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality.
* Has known history of Guillain-Barré Syndrome.
* Has clinical signs of active infection and/or an oral temperature of greater than or equal to 38°C (100.4°F). Study entry may be deferred for such individuals at the discretion of the Principal Investigator (PI).
* Has history of neurological disorders or seizures, with exception of a single febrile seizure during childhood.
* Has confirmed or suspected immunosuppressive condition (including cancer), or a previously diagnosed immunodeficiency disorder (congenital or acquired).
* Currently receiving (within the 90 days before receiving the study vaccines) immunosuppressive or immunomodulative therapy, systemic corticosteroids, and including the following medications:
* Chronic or long-term corticosteroids: greater than 15mg/day of oral prednisolone or equivalent daily;
* Sporadic corticosteroids: greater than 40mg/day of oral prednisolone or equivalent for more than 2 courses of greater than 14 days in the 3 months preceding vaccination;
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.

Note: Use of topical or inhalant corticosteroids prior to administration of the study vaccines or throughout the study is acceptable.

* Participated in a clinical trial or use of an investigational compound within 30 days before receiving the study vaccine or plans to enter a study during the study period.
* Was vaccinated with a registered vaccine within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to receiving the study vaccine.
* Currently treated with cytotoxic drugs or at any time during the 6 months before administration of the study vaccines.
* Has major congenital defects or serious chronic illness.
* Has evidence or history of (within the previous 12 months) drug or alcohol abuse.
* Is unwilling or unable to comply with the study protocol.
* Has a history of psychiatric disorders that, in the opinion of the PI, would prevent the subject from giving proper informed consent or otherwise interfere with the study.
* Is a resident of nursing home or long-term care facility.
* Has any condition that, in the opinion of the PI, would prevent the subject from complying with all aspects of the protocol or will put the subject at unnecessary risk.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1359 (Actual)
Dates: Start 2006-06; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Immunogenicity endpoints of seroprotection rate and seroconversion rate will be assessed. | Day 0 prior to vaccination and day 21 after vaccination.

SECONDARY OUTCOMES:
Comparison of the geometric mean titers to influenza hemagglutinin antigens after vaccination of the active treatment arms. | Day 0 prior to vaccination and day 21 after vaccination.
The number and rate of the type, frequency and intensity of adverse events in the active treatment arms. | Solicited adverse events through day 4 (days 0, 1, 2, 3, 4) following vaccination; unsolicited adverse events to day 21 after vaccination.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Stanford University, Stanford, California
  - University of Iowa, Iowa City, Iowa
  - University of Maryland Baltimore, Baltimore, Maryland
  - Saint Louis University, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Clinical Alliance for Research & Education - Infectious Diseases, Annandale, Virginia

REFERENCES:
- [Background] Talbot HK, Keitel W, Cate TR, Treanor J, Campbell J, Brady RC, Graham I, Dekker CL, Ho D, Winokur P, Walter E, Bennet J, Formica N, Hartel G, Skeljo M, Edwards KM. Immunogenicity, safety and consistency of new trivalent inactivated influenza vaccine. Vaccine. 2008 Jul 29;26(32):4057-61. doi: 10.1016/j.vaccine.2008.05.024. Epub 2008 Jun 2. PMID 18602726